CLINICAL TRIAL: NCT06774924
Title: "Clinical Ultrasound, a New Link Between Town and Hospital in Seine-Saint-Denis". (ECHO93)
Acronym: ECHO93
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP 240421; N° IDRCB: 2024-A (Other: ANSM)
Record Dates: First submitted 2024-10-18; First posted 2025-01-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Diagnosis; Clinical Ultrasound
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- echoscopy examination using the echOpen probe (Other): In addition to standard care, each patient will have a systematic 4-point echoscopy examination using the echOpen probe: liver, spleen, lymph nodes, thyroid and, depending on symptoms, lung, kidney, bladder, abdomen.
  The echOpen probe is CE marked. It will be used for all indications except certain areas of the body (thyroid, lymph nodes, bladder, liver, spleen, kidney, bladder and lymph nodes).
  Interventions: Device: Echoscopy examination using the echOpen probe

INTERVENTIONS:
Device: Echoscopy examination using the echOpen probe — In addition to standard care, each patient will have a systematic 4-point echoscopy examination using the echOpen probe: liver, spleen, lymph nodes, thyroid and, depending on symptoms, lung, kidney, bladder, abdomen.
  The echOpen probe is CE marked. It will be used for all indications except certain areas of the body (thyroid, lymph nodes, bladder, liver, spleen, kidney, bladder and lymph nodes).
  In addition to echoscopy with the echOpen probe, patient and physician satisfaction questionnaires will be used as part of this study.
  Other Names: patient and investigator satisfaction questionnaires

SUMMARY:
The ECHO93 study is a non-healthcare interventional study. Its aim is to evaluate the effect of introducing the echOpen probe into the management of patients referred to the Jean Verdier UDR, in terms of time to diagnosis.

The study is divided into 3 phases:

Phase 1: opening of the Rapid Diagnosis Unit (UDR) at Jean Verdier Hospital Phase 2: Opening of the Jean Verdier Hospital UDR, MSP Pantin, Dr TAYBALY's medical practice in Aulnay-sous-Bois, one month after the start of phase 1.

Phase 3: Opening of the Jean Verdier Hospital Health Bus, one month after the start of phase 2.

DETAILED DESCRIPTION:
This research will be carried out in 3 phases:

* Phase 1: implementation of the tool within the hospital for UDR doctors and evaluation of the effect of this implementation on the organizations: shorter time to diagnosis, increased accuracy of diagnosis, reduced number of complementary examinations. This first phase will begin with EchOpen training for doctors, and will continue with inclusions and testing of the added value of using the probe within the UDR.
* Phase 2: implementation of the tool in the structures referring patients to the UDR, whether the SAU de Jean Verdier, for clearing before referral to the UDR, or the structures of town doctors (CPTS Livry Gargan, MSP Pantin and Cabinet Médical du Dr TAYBALY at Aulnay-sous-Bois) for clearing before referral to the UDR. As in phase 1, the aim is to assess the effect of the new approach on organization, and to report on follow-up indicators, such as the number of patients with direct access to biopsy, the reduction in diagnosis time, and the targeting and reduction of additional examinations. This second phase will begin one month after phase 1, starting with EchOpen training for doctors and continuing with inclusions and experimentation within the adult emergency departments of Jean Verdier Hospital and the multi-professional health centers named above.
* Phase 3: implementation of the tool in the Health Bus, as part of the "go-to" approach. The monitoring indicator will be the number of situations in which the echOpen solution has made it possible to sort between pathologies that require an emergency service or that can be managed in the Health Bus. This third phase will begin one month after phase 2, starting with EchOpen training for doctors and continuing with inclusions and testing of the probe in the Health Bus.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient over 18 years of age
2. Patient with signed informed consent
3. Patient managed by:

   * one of the structures involved (UDR/ SAU Jean Verdier, MSP Pantin, Cabinet Médical du Dr TAYBALY à Aulnay-sous-Bois) for referral to the UDR for rapid diagnosis (phases 1 and 2)
   * the Health Bus (phase 3)

Exclusion Criteria:

1. Patient on the UDR iron-deficiency anemia clinical pathway
2. Patient deprived of liberty by judicial or administrative decision
3. Patient who does not speak French and cannot benefit from the presence of a relative or translator (physical or online)
4. Patient with a contraindication to the use of EchOPen:

   * patients with a body mass index greater than 34.9 kg/m2
   * life-threatening patients requiring emergency medical care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of introducing the echOpen probe into the management of patients referred to the Jean Verdier Rapid Diagnostic Unit (UDR) on time to diagnosis. | Visite discharge from the RDU ( Maximum 2 months after inclusion visit)
  The time between the first contact with the Rapid Diagnosis Unit (RDU) and the date of the diagnosis (date of discharge from the RDU) in patients who had an ultrasound scan with the echOpen probe in consultation at the RDU (phase 1) and in patients who had it in consultation with a general practitioner or in the emergency department (phase 2), compared with the time before the echOpen was introduced.

SECONDARY OUTCOMES:
Evaluate the effect of introducing the echOpen probe in the management of patients referred to the Jean Verdier UDR on time to diagnosis according to where the tool is used. | Visite discharge from the RDU ( Maximum 2 months after inclusion visit)
  - The number of complementary examinations prescribed/avoided, in comparison with the number of examinations prior to the introduction of the echOpen.
Evaluate the effect of introducing the echOpen probe in the management of patients referred to the Jean Verdier UDR on time to diagnosis according to where the tool is used. | Visite discharge from the RDU ( Maximum 2 months after inclusion visit)
  - The time between the first consultation and the radioguided biopsy, if this is to be carried out
Evaluate the effect of introducing the echOpen probe in the management of patients referred to the Jean Verdier UDR on time to diagnosis according to where the tool is used. | Visite discharge from the RDU ( Maximum 2 months after inclusion visit)
  - The number of patients accessing the UDR day hospital directly will be evaluated in patients having had an echoscopy with the echOpen probe in consultation at the UDR (phase 1) in comparison with the number of patients before the introduction of the echOpen.
Evaluate the effect of introducing the echOpen probe in the management of patients referred to the Jean Verdier UDR on time to diagnosis according to where the tool is used. | Visite discharge from the RDU ( Maximum 2 months after inclusion visit)
  - The number of patients referred to the emergency department facilitated by the echOpen probe will be evaluated among patients who had an echOpen probe in the Health Bus (phase 3), compared with the number of patients before the echOpen was introduced.
Evaluate the satisfaction of physicians participating in the study with the introduction of the echOpen probe in the management of patients referred to the Jean Verdier UDR. | Through study completion, an average of 2 years for phase 1 and 2, at each inclusion visit of patient (day 1) for phase 3
  Physician satisfaction (phases 1 and 2) will be assessed by a questionnaire carried out at the end of the study. For Health Bus doctors (phase 3), the questionnaire will be completed after each patient consultation. A visual analog scale will be proposed in this questionnaire to assess doctors' overall satisfaction with the use of EchOpen. This scale ranges from 0 (very dissatisfied) to 10 (very satisfied).
Evaluate the satisfaction of physicians participating in the study with the introduction of the echOpen probe in the management of patients referred to the Jean Verdier UDR. | once a week throughout the entire inclusion period which is 16 months
  Physicians' satisfaction will also be assessed by a weekly questionnaire sent directly to them by the EchOpen team.
To assess patient satisfaction with the introduction of the echOpen probe in the management of patients referred to the Jean Verdier UDR. | Visit discharge from the RDU ( Maximum 2 months after inclusion visit) for pahse 1 and 2. At the Inclusion visit (day 1) for phase 3
  Patient satisfaction (phases 1 and 2) will be assessed by a questionnaire administered on discharge from the UDR. For Health Bus patients (phase 3), the questionnaire will be carried out at the Inclusion/Final visit. This questionnaire will include a visual analog scale to assess patients' overall satisfaction with the EchOpen. The scale ranges from 0 (very dissatisfied) to 10 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Anne BOURGARIT, PUPH, Study Director — HUPSSD
Locations (1):
- Unite de Diagnostic Rapide - Medecine Interne Hopital Jean Verdier, Bondy, France